CLINICAL TRIAL: NCT07230990
Title: Mechanisms Of Orbitofrontal Stimulation in Depression (MOOD)
Brief Title: Mechanisms Of Orbitofrontal Stimulation in Depression
Acronym: MOOD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Subha Subramanian (Other)
Responsible Party: Sponsor-Investigator, Subha Subramanian, Instructor of Psychiatry, TMS Director, Harvard University Faculty of Medicine
Organization: Harvard University Faculty of Medicine (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025P000673
Record Dates: First submitted 2025-11-06; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Depression; Transcranial magnetic stimulation (TMS); orbitofrontal cortex; Frontal pole
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into active or sham TMS groups and active or sham TMS to the right OFC. They will then undergo a washout period. After this, all participants will receive active TMS to the OFC. This region corresponds to the FP2 electrode location in the international 10-20 EEG system and is also referred to as the frontal pole.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, investigators, and outcome assessors will be blinded to treatment allocation (active vs. sham TMS). Blinding will be maintained using coded assignments that indicate which side of the MagPro Cool B65 A/P coil (MagVenture A/S, Denmark) is positioned for stimulation. This procedure ensures that all study personnel remain unaware of stimulation condition throughout the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active OFC stimulation (Active Comparator): Continuous intermittent theta burst stimulation (cTBS, a type of inhibitory TMS) to the right OFC.
  Interventions: Device: Active TMS
- Sham OFC stimulation (Sham Comparator): Sham TMS treatment to the right OFC
  Interventions: Device: Sham TMS

INTERVENTIONS:
Device: Sham TMS — The MagVenture MagPro system's active/sham coil (e.g., Cool-B65 A/P) will be used to deliver either active or sham TMS. The sham mode reproduces the same clicking sound and scalp sensation as active stimulation but does not induce cortical activation. The built-in MagPro double-blind feature ensures operator, participant, and investigator blinding. All participants will be randomized to receive active or sham TMS to the OFC in the first phase.
  Arms: Sham OFC stimulation
Device: Active TMS — TMS uses magnetic fields generated by a coil placed next to the scalp to alter brain activity at a specific region (i.e., OFC) protocol. Here, active TMS protocol is continuous intermittent theta burst stimulation (cTBS, a type of inhibitory TMS) to the right OFC. Investigators will use the MagVenture MagPro system's active/sham coil (e.g., Cool-B65 A/P) to deliver either active or sham TMS. All participants will be randomized to receive active or sham TMS to the OFC in the first phase. In the second phase, all participants will receive active TMS to the OFC. The active protocol to the right OFC is: continuous intermittent theta burst stimulation (cTBS, a type of inhibitory TMS).
  Arms: Active OFC stimulation

SUMMARY:
The orbitofrontal cortex (OFC), a region involved in emotional regulation, decision making, and reward processing, is a key area linked to antidepressant response. This study tests whether noninvasive stimulation of the OFC using transcranial magnetic stimulation (TMS) can improve depressive symptoms. TMS uses magnetic fields generated by a coil placed next to the scalp to alter brain activity.

DETAILED DESCRIPTION:
The main purpose of this study is to test a new treatment target for major depressive disorder (MDD) and to understand the brain mechanisms that may lead to antidepressant response. The treatment target of this study is the right orbitofrontal cortex (OFC), a brain region towards the front of the brain involved in emotion regulation, reward-processing, and decision-making. Other studies have shown that stimulating the OFC can improve depression symptoms. However, no study has yet directly compared the effects of real (active) versus placebo (sham) OFC stimulation on both mood and brain function. Comparison of active versus sham treatment is key in medical research. This study aims to fill that gap by comparing active versus sham stimulation of the right OFC in people with MDD who are currently experiencing moderate to severe symptoms. Participants will take part in a two phases: a triple-blind, randomized, sham-controlled phase, followed by an open-label phase where all participants receive active OFC stimulation.

Aim 1:

To determine whether active TMS targeting the right OFC, compared to sham stimulation at the same site, reduces depressive symptom severity in individuals with MDD.

Aim 2:

To test whether active TMS to the right OFC, compared to sham stimulation at the same site, reduces ruminative symptoms in individuals with MDD.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Must be able to read, speak and understand English
* DSM-5 diagnosis of major depressive disorder, experiencing a moderate to severe depressive episode (Hamilton Depression Rating Scale score greater than or equal to 17 points)
* Must be judged by study staff to be capable of completing the study procedures
* Participants will be in stable outpatient treatment with no recent (within the past 30 days) hospitalizations or changes in their medication regimens

Exclusion Criteria:

* DSM-5 moderate to severe substance use disorder within the past three months, based on Structured Clinical Interview for DSM-5
* Conditions that might result in increased risks of side effects or complications from rTMS or MRI, including:

  * History of fainting spells of unknown or undetermined etiology that might constitute seizures
  * Diagnosis of epilepsy with the exception of a single seizure of benign etiology (e.g., febrile seizures) in the judgment of a board-certified neurologist
  * Current or past history of a neurological disorder, such as stroke, a progressive neurologic disease, or intracranial brain lesion(s); and history of previous neurosurgery or head trauma that resulted in residual neurologic impairment
  * Any unstable medical condition
  * Any metal in the brain or skull (excluding dental fillings) unless cleared by the responsible covering MD
  * Any devices which could be affected by TMS or MRI such as a pacemaker, medication pump, nerve stimulator, cochlear implant, TENS unit, ventriculo-peritoneal shunt unless cleared by the responsible covering MD
  * Pregnancy; All female participants will be required to have a pregnancy test; any participant who is pregnant will not be enrolled in the study. The pregnancy test will be administered by study staff trained to administer point of care pregnancy testing that complies with institutional laboratory policies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory II (BDI-II) | The survey will be administered at 4 timepoints: Day 1 (baseline) and Day 10 (last day) of randomized phase; Day 1 (baseline) and Day 10 (last day) of open-label phase.
  The BDI-II is a 21-item self-report questionnaire assessing the severity of depressive symptoms over the past two weeks. Each item is rated from 0 to 3, reflecting increasing symptom severity. The total score range is 0 to 63 points, where higher scores indicate worse depressive symptoms. The investigators will examine the change in BDI-II scores in each experimental phase (randomized and open-label).
Hamilton Depression Rating Scale (HDRS) - 24 item version | The survey will be administered at 4 timepoints: Day 1 (baseline) and Day 10 (last day) of randomized phase; Day 1 (baseline) and Day 10 (last day) of open-label phase.
  The HDRS is a clinician-rated scale assessing the severity of depressive symptoms across mood, somatic, and cognitive domains. Items are scored on either 3- or 5-point scales depending on the symptom. The score ranges from 0 to 76, with higher scores reflecting greater severity.
Rumination Response Scale (RRS) | The survey will be administered at 4 timepoints: Day 1 (baseline) and Day 10 (last day) of randomized phase; Day 1 (baseline) and Day 10 (last day) of open-label phase.
  The RRS is a 22-item self-report questionnaire measuring the tendency to engage in repetitive, negative thinking about one's distress or mood. Each item is rated from 1 ("almost never") to 4 ("almost always"). Scores range from 22 to 88 points, with higher scores indicating greater rumination.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stolinsky DC. Asklepios. Ann Intern Med. 1996 Aug 1;125(3):253-4. doi: 10.7326/0003-4819-125-3-199608010-00021. No abstract available. PMID 8686990
- [Result] Hanlon CA, Dowdle LT, Correia B, Mithoefer O, Kearney-Ramos T, Lench D, Griffin M, Anton RF, George MS. Left frontal pole theta burst stimulation decreases orbitofrontal and insula activity in cocaine users and alcohol users. Drug Alcohol Depend. 2017 Sep 1;178:310-317. doi: 10.1016/j.drugalcdep.2017.03.039. Epub 2017 May 30. PMID 28686990
- [Result] Cui H, Ding H, Hu L, Zhao Y, Shu Y, Voon V. A novel dual-site OFC-dlPFC accelerated repetitive transcranial magnetic stimulation for depression: a pilot randomized controlled study. Psychol Med. 2024 Oct 23;54(14):1-14. doi: 10.1017/S0033291724002289. Online ahead of print. PMID 39440449
- [Result] Kringelbach ML. The human orbitofrontal cortex: linking reward to hedonic experience. Nat Rev Neurosci. 2005 Sep;6(9):691-702. doi: 10.1038/nrn1747. PMID 16136173
- [Result] Fettes P, Schulze L, Downar J. Cortico-Striatal-Thalamic Loop Circuits of the Orbitofrontal Cortex: Promising Therapeutic Targets in Psychiatric Illness. Front Syst Neurosci. 2017 Apr 27;11:25. doi: 10.3389/fnsys.2017.00025. eCollection 2017. PMID 28496402
- [Result] Tadayonnejad R, Citrenbaum C, Ngo TDP, Corlier J, Wilke SA, Slan A, Distler MG, Hoftman G, Adelekun AE, Leuchter MK, Koek RJ, Ginder ND, Krantz D, Artin H, Strouse T, Bari AA, Leuchter AF. Right lateral orbitofrontal cortex inhibitory transcranial magnetic stimulation for treatment of refractory mood and depression. Brain Stimul. 2023 Sep-Oct;16(5):1374-1376. doi: 10.1016/j.brs.2023.09.011. Epub 2023 Sep 15. No abstract available. PMID 37716637
- [Result] Prentice A, Kolken Y, Tuttle C, van Neijenhof J, Pitch R, van Oostrom I, Kruiver V, Downar J, Sack AT, Arns M, van der Vinne N. 1Hz right orbitofrontal TMS benefits depressed patients unresponsive to dorsolateral prefrontal cortex TMS. Brain Stimul. 2023 Nov-Dec;16(6):1572-1575. doi: 10.1016/j.brs.2023.10.005. Epub 2023 Oct 13. No abstract available. PMID 37839775
- [Result] Feffer K, Fettes P, Giacobbe P, Daskalakis ZJ, Blumberger DM, Downar J. 1Hz rTMS of the right orbitofrontal cortex for major depression: Safety, tolerability and clinical outcomes. Eur Neuropsychopharmacol. 2018 Jan;28(1):109-117. doi: 10.1016/j.euroneuro.2017.11.011. Epub 2017 Nov 17. PMID 29153927
- [Result] Rao VR, Sellers KK, Wallace DL, Lee MB, Bijanzadeh M, Sani OG, Yang Y, Shanechi MM, Dawes HE, Chang EF. Direct Electrical Stimulation of Lateral Orbitofrontal Cortex Acutely Improves Mood in Individuals with Symptoms of Depression. Curr Biol. 2018 Dec 17;28(24):3893-3902.e4. doi: 10.1016/j.cub.2018.10.026. Epub 2018 Nov 29. PMID 30503621